CLINICAL TRIAL: NCT01378507
Title: Endoscopic Submucosal Dissection for Gastrointestinal Neoplasms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Lu Zhong-Sheng, Department of Gastroenterology and Hepatology
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20110526004
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-05

CONDITIONS: Digestive System Diseases
Keywords: endoscopic submucosal dissection; gastrointestinal neoplasm
MeSH Terms: conditions — Digestive System Diseases; Gastrointestinal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endoscopic Submucosal Dissection (Experimental): Single-arm for ESD procedure and retrospective surgical procedure(Laparoscopy, Open surgery)data collection
  Interventions: Behavioral: endoscopic submucosal dissection

INTERVENTIONS:
Behavioral: endoscopic submucosal dissection — ESD was carried out by using a single-channel upper gastrointestinal endoscope with a water-jet system (Q260J; Olympus Optical Co, Tokyo, Japan) and a high-frequency generator with an automatically controlled system (ENDOCUT mode) (Erbotom ICC 200; ERBE Elektromedizin GmbH, Tübingen, Germany). The transparent attachment was fitted on the tip of the endoscope mainly to obtain a constant endoscopic view and to create tension on the connective tissue for the submucosal dissection.
  Other Names: Endoscopic Submucosal Dissection(ESD)

SUMMARY:
Endoscopic submucosal dissection (ESD) is a newly developed technique in the field of endoscopic treatment for GI neoplasms, because of its high rate of en bloc resection. The purpose of this study is to evaluate the efficacy and safety of ESD for GI neoplasms.

DETAILED DESCRIPTION:
Endoscopic mucosal resection (EMR) is widely accepted as a minimally invasive treatment for GI neoplasms.However, one disadvantage of EMR is that lesions larger than 2 cm in diameter must be removed in pieces, which may result in a high recurrence rate of residual tumor tissue. In addition, in most patients, pathological assessment cannot be conducted after the procedure. ESD can overcome the disadvantages of EMR. However, it is difficult to perform ESD for GI neoplasms because of the high rate of complications.

ELIGIBILITY:
Inclusion Criteria:

* Submucosal tumor
* Mucosal tumor (T1) in patients unsuitable for surgery

Exclusion Criteria:

* Endoscopic ultrasound (EUS) or CT signs of metastasis
* Insufficient access to tumor

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-06 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
The lesion result before ESD | within 7 days before ESD
  Including the location, morphology and size under endoscopy and narrow banding image of lesion.
Short-term result after ESD | whithin 7 days after ESD
  Including en bloc and curative resection rate, the specimen size, complications, lateral and vertical margin exposure of tumor, and lymphatic or vascular invasion.

SECONDARY OUTCOMES:
The safety of ESD procedure | 3months, 6months, 1year, 2years, 3years, 4years and 5years after ESD
  including the endoscopic examination at 3months, 6months, 1year, 2years, 3years, 4years and 5years after ESD

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-Sheng Lu, M.D., Study Chair — Chinese PLA General Hospital; Yun-Sheng Yang, M.D., Study Director — Chinese PLA General Hospital; Jin Huang, M.D., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Huang J, Yang YS, Lu ZS, Wang SF, Yang J, Yuan J. Detection of superficial esophageal squamous cell neoplasia by chromoendoscopy-guided confocal laser endomicroscopy. World J Gastroenterol. 2015 Jun 14;21(22):6974-81. doi: 10.3748/wjg.v21.i22.6974. PMID 26078575